CLINICAL TRIAL: NCT05448885
Title: Neoadjuvant Chemotherapy Plus Tislelizumab Followed by Concurrent Chemoradiotherapy and Maintenance Therapy With Tislelizumab in Patients With Stage IVA Nasopharyngeal Carcinoma: A Single-arm, Phase II Trial
Brief Title: Neoadjuvant and Adjuvant Tislelizumab for Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Yi Junlin, chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21/273-2944
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — tislelizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: GP combined with Tislelizumab neoadjuvant therapy+CCRT+Tislelizumab adjuvant therapy (Experimental): Patients receive neoadjuvant therapy with gemcitabine(1000mg per square meter on day 1,8) , cisplatin (25mg per square meter on day 1-3) and tislelizumab(200mg) every three weeks for 2 cycles before radiotherapy, then followed by concurrent IMRT and cisplatin (100mg per square meter) concurrent every three weeks during radiotherapy ,then followed by adjuvant therapy with tislelizumab(200mg) every three weeks for 13 cycles after radiotherapy
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Patients receive neoadjuvant therapy with gemcitabine(1000mg per square meter on day 1,8) , cisplatin (25mg per square meter on day 1-3) and tislelizumab(200mg) every three weeks for 2 cycles before radiotherapy, then followed by concurrent IMRT and cisplatin (100mg per square meter) concurrent every three weeks during radiotherapy ,then followed by adjuvant therapy with tislelizumab(200mg) every three weeks for 13 cycles after radiotherapy
  Other Names: gemcitabine, cisplatin

SUMMARY:
To estimate the efficacy and safety of tislelizumab for stage IVA locally advanced nasopharyngeal carcinoma combined with induction chemotherapy and concurrent chemoradiotherapy, followed by maintenance therapy

DETAILED DESCRIPTION:
Platinum-based concurrent chemoradiotherapy is the standard of care for patients with locoregionally advanced nasopharyngeal carcinoma(NPC). Gemcitabine plus cisplatin(GP) has been demonstrated an effective chemotherapy regimen for NPC patients in previous studies. The results of GP combined with concurrent chemoradiotherapy in the treatment of locoregionally advanced nasopharyngeal carcinoma showed 10% of locoregionally advanced NPC patients had complete response after three cycles of GP neoadjuvant chemotherapy, and GP neoadjuvant chemotherapy added to chemoradiotherapy significantly improved recurrence-free survival (85.3% vs 76.5%) and overall survival (94.6% vs 90.3%) among locoregionally advanced NPC patients , as compared with chemoradiotherapy alone. Therefore, GP regimen has been established as the highest level of evidence-based neoadjuvant chemotherapy in the 2020 National Comprehensive Cancer Network (NCCN) guidelines. Recently, immune checkpoint inhibitors, such as anti-programmed cell death-1 (PD-1)monoclonal antibody has shown promising efficacy in the treatment of tumor patients. Clinical trials have shown objective response rates of 20.5%-34% in patients with recurrent or metastatic NPC patients receiving anti PD-1 monoclonal antibody immunotherapy including pembrolizumab, nivolumab, camrelizumab, and toripalimab. The current NCCN guidelines recommend anti PD-1 monoclonal antibody as a second-line treatment for recurrent or metastatic NPC. More and more evidence show that immunotherapy combined with chemotherapy has a synergistic effect in treating tumors. GP chemotherapy combined with anti PD-1 antibody has achieved the initial effect in NPC. Phase 1 trials have shown the combination of camrelizumab plus GP chemotherapy in recurrent or metastatic NPC led to a proportion of 91% patients achieving an objective response. In addition, previous studeis showed that PD-1 antibody adjuvant therapy had good feasibility and effectiveness in the treatment of nasopharyngeal carcinoma. Tislelizumab, approved by the National Medical Products Administration in China, is an anti-PD-1 monoclonal IgG4 antibody with higher affinity to PD-1 than pembrolizumab and nivolumab and was engineered to minimize binding to FcγR on macrophages in order to abrogate antibody-dependent phagocytosis, a mechanism of T-cell clearance and potential resistance to anti-PD-1 therapy. Multiple clinical trials have shown strong anti-neoplastic activity of tislelizumab in various tumors including NPC. Clinical trial has shown an objective response rates of 43% in patients with recurrent metastatic nasopharyngeal carcinoma treated with tirelizumab, which is superior to other anti PD-1 monoclonal antibodys. So we hypothesize that GP neoadjuvant chemotherapy combined with tislelizumab and tislelizumab adjuvant therapy could further improve survival of patients with locaregionally advanced NPC. Based on this, this study aims to evaluate the efficacy and safety of gemcitabine plus cisplatin chemotherapy combined with tislelizumab neoadjuvant therapy, followed by cisplatin based concurrent chemoradiotherapy, then followed by tislelizumab adjuvant therapy in the patients with locoregionally advanced nasopharyngeal carcinoma, to provide new evidence for individualized comprehensive treatment in NPC.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects are not limited by gender, age from 18 to 70 years old;
2. Histopathologically confirmed non-keratinizing squamous cell carcinoma of the nasopharynx;
3. Locally advanced nasopharyngeal squamous cell carcinoma diagnosed as T4 or N3 stage according to AJCC 8th edition staging;
4. ECOG score 0-1;
5. without distant metastasis;
6. This treatment must be the first course of treatment, and has not received any anti-tumor treatment such as radiotherapy and chemotherapy, immune or biological therapy in the past.
7. The expected survival is expected to be no less than 6 months.
8. No contraindications to chemotherapy, immunotherapy and radiotherapy;

Exclusion Criteria:

1. Received any systemic anti-tumor therapy for target lesions in the past;
2. Previously experienced head and neck radiation therapy;
3. Those who have received any immunotherapy such as anti-PD-1/PD-L1 monoclonal antibody, anti-CTLA-4 monoclonal antibody in the past;
4. Subjects who have been vaccinated with anti-tumor vaccines or other drugs with immunomodulatory functions (such as interleukin-2, thymosin, lentinan, etc.) within 1 month before enrollment, or who will be vaccinated with live attenuated vaccines. subject;
5. Subjects who have used corticosteroids (>10 mg/day prednisone or other equivalent hormones) or other immunosuppressive agents for systemic treatment within 1 month before enrollment. In the absence of active autoimmune disease, inhaled or topical corticosteroids and adrenal hormone replacement therapy at therapeutic doses of prednisone ≤10 mg/day are permitted;
6. Patients with pleural effusion, pericardial effusion or ascites that need to be drained with clinical symptoms, or who have received serous cavity effusion drainage for the purpose of treatment within 2 weeks before enrollment;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
2-y PFS | 2 years
  defined as the time from random assignment to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first after 2 years of treatment.

SECONDARY OUTCOMES:
CR | 1 year
  CR assessed by investigator, according to the Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI). Disease response evaluated after the completion of the neoadjuvant therapy. Complete response defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging (MRI) .
OS | 3 years
  defined as the time from random assignment to death from any cause or censored at the date of last follow-up.
PFS | 3 years
  defined as the time from random assignment to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first.
safety | 3 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events (acute toxicity) and late radiation toxicities were assessed by NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center /National Clinical Research Center for Cancer/Cancer Hospital, CAMS & PUMC, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No